CLINICAL TRIAL: NCT03230630
Title: Early-morning Plasma Melatonin Levels Predict Cardiovascular Mortality After Acute Myocardial Infarction
Brief Title: Plasma Melatonin AND Mortality After Acute Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Li Jing Wei, Doctor, Chinese PLA General Hospital
Other Study IDs: melatonin-AMI
Record Dates: First submitted 2017-07-24; First posted 2017-07-26 (Actual); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Melatonin; Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: plasma melatonin levels

SUMMARY:
Pre-clinical and clinical studies have demonstrated that melatonin has cardio-protection effects. Melatonin has anti-inflammatory, antioxidant, antihypertensive, antithrombotic and antilipaemic properties, which plays important roles in a variety of cardiovascular pathophysiologic processes. Nocturnal melatonin levels decreased after AMI, and lower serum melatonin concentrations after AMI are associated with more heart failure and cardiac death and left ventricular remodeling. Moreover in women with increased BMI, lower melatonin secretion is associated with higher risks of MI. Early-morning blood collection is easier in clinical practice. Therefore, the investigators carried out a cohort study to evaluate the prognostic value of plasma soluble melatonin in hospitalized patients with acute myocardial infarction (AMI).

ELIGIBILITY:
Inclusion Criteria:

* consecutive patients of acute AMI come to department of cardiology, 301 hospital (Beijing, China),absent of cardiogenic shock, and survival for at least 24 h after percutaneous coronary intervention treatment.

Exclusion Criteria:

* patients with autoimmune diseases, collagen tissue diseases, drug addiction, radiotherapy, patients receiving immunosuppressive treatment, taking sedatives, antiepileptic drugs, tricyclic antidepressants or any medication known to influence melatonin metabolism, psychiatric sleeping disorders, shift workers, and subjects with jet-lag syndrome

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A single center study on PCI-treated myocardial infarction patients
Sampling Method: Non-Probability Sample
Enrollment: 732 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2015-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
cardiovascular mortality | The median follow-up was 31.6 months

SECONDARY OUTCOMES:
non-cardiovascular mortality | The median follow-up was 31.6 months
Myocardial infarction | The median follow-up was 31.6 months
heart failure readmission | The median follow-up was 31.6 months
  readmission to any hospital due to diagnosed heart failure
Stroke | The median follow-up was 31.6 months
  defined using the World Health Organization criteria